CLINICAL TRIAL: NCT03473977
Title: A Randomized, Double-Blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy of Benralizumab (Anti-IL5RA) in Subjects With Eosinophilic Gastritis
Brief Title: Benralizumab for Eosinophilic Gastritis (BEGS)
Acronym: BEGS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-1701
Record Dates: First submitted 2018-02-28; First posted 2018-03-22 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Eosinophilic Gastritis or Gastroenteritis
MeSH Terms: conditions — Eosinophilic enteropathy; Gastroenteritis | interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: Participants will receive doses of drug or placebo. Optional open label extensions available following the double blind period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant/care providers, investigators, and outcome assessor (pathology) were blinded to assignment. Randomization performed by external investigational pharmacy staff (dispenses the drug/placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab (Experimental): Subcutaneous dose of 30 mg of Benralizumab every 4 weeks
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Subcutaneous dose of Placebo every 4 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab (anti-IL5Ra) will be injected every 4 weeks in doses of 30 mg (total of 3 injections) in subjects with active Eosinophilic Gastritis.
  Other Names: Fasenra
  Arms: Benralizumab
Biological: Placebo — Placebo will be injected every 4 weeks (total of 3 injections) as a comparator to Benralizumab in subjects with active Eosinophilic Gastritis.
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy of Benralizumab (Anti-IL5RA) in Subjects With Eosinophilic Gastritis.

DETAILED DESCRIPTION:
Primary Objective:

To assess the efficacy of repeat subcutaneous (SC) doses of benralizumab, compared with placebo, to reduce eosinophilic inflammation in the gastrointestinal tract of patients with Eosinophilic Gastritis

Secondary Objectives:

To assess changes in endoscopic score, histological features, blood and biopsy eosinophil counts, clinical symptoms, and gastric tissue transcriptome before and after treatment with benralizumab.

26 subjects are planned to be enrolled into the study at Cincinnati Children's Hospital Medical Center. Qualifying Subjects will receive subcutaneous injections every 4 weeks (3 total) of benralizumab/Placebo, followed by optional Open Label Extension periods.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Males and females between the ages of 12-60 years with confirmed diagnosis of EG involving stomach; involvement of eosinophilic inflammation in other gastrointestinal segments will be allowed but not required or sufficient.
* Histologically active EG at time of screening, with a peak Gastric count of ≥ 30 eos/hpf in at least 5 hpfs.
* Must be symptomatic (defined as having experienced symptoms within 4 weeks prior to enrollment).
* Blood eosinophilia (defined as having an absolute eosinophil count > 500 cells per microliter of blood) at least once during the 6 months prior to enrollment.
* Must be on baseline anti-eosinophilic gastritis/eosinophilic gastroenteritis therapy as long as there is agreement to not change their dosage unless medically indicated; OR, must have failed anti-eosinophilic gastritis/eosinophilic gastroenteritis in the past, including diet therapy.
* Clinical symptoms (i.e., abdominal pain, bloating, vomiting, diarrhea) severe enough to impact daily life (e.g., school/work attendance, social activities) ≥ 2 days/week for 3 of the 4 weeks prior to enrollment despite treatment (such as diet, proton pump inhibitors or corticosteroids).
* Female subjects: Women of childbearing potential (WOCBP) must use an effective form of birth control (confirmed by the Investigator). Effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective intrauterine device/ levonogestrel Intrauterine system, Depo-Provera(tm) injections, oral contraceptive, and Evra Patch(tm) or Nuvaring(tm). WOCBP must agree to use effective method of birth control, as defined above, from enrollment, throughout the study duration and within 16 weeks after last dose of investigational product, and have negative serum pregnancy test result on Visit 1.
* Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of visit -1 without an alternative medical cause. The following age-specific requirements apply:
* Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.
* Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
* All male subjects who are sexually active must agree to use an acceptable method of contraception (condom with or without spermicide, vasectomy) from Visit 1 until 16 weeks after their last dose.

Exclusion Criteria:

* Concurrent H. pylori gastritis or parasitic infection
* Other gastrointestinal disorders such as Crohn's disease, inflammatory bowel disease, or Celiac disease, eosinophilic granulomatosis with polyangiitis (EGPA), drug hypersensitivity or connective tissue rheumatological disorders,
* Esophageal stricture that prevents the easy passage of a standard endoscope
* Use of any investigational biologic drug within 6 months prior to screening
* Hypereosinophilic syndrome, defined by multiple organ involvement (with the exception of atopic disease or EGID) and persistent blood absolute eosinophil count ≥1500/mcL.
* History of cancer: Subjects who have had basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to the date informed consent, and assent when applicable was obtained. Subjects who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to the date informed consent, and assent when applicable, was obtained.
* A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy.
* Pregnant or nursing
* Receipt of any investigational non-biologic within 30 days or 5 half-lives prior to visit 1, whichever is longer.
* A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.
* Any other medical illness that precludes study involvement
* Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to be enrolled.
* Patients who are currently receiving or have previously received benralizumab or any other type of anti-interleukin therapy (i.e. mepolizumab, reslizumab, lebrikizumab etc.) within the last 6 months or 5 half-lives whichever is longer.
* History of anaphylaxis to any biologic therapy or vaccine.
* Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2022-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Rothenberg, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kliewer KL, Murray-Petzold C, Collins MH, Abonia JP, Bolton SM, DiTommaso LA, Martin LJ, Zhang X, Mukkada VA, Putnam PE, Kellner ES, Devonshire AL, Schwartz JT, Kunnathur VA, Rosenberg CE, Lyles JL, Shoda T, Klion AD, Rothenberg ME. Benralizumab for eosinophilic gastritis: a single-site, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Gastroenterol Hepatol. 2023 Sep;8(9):803-815. doi: 10.1016/S2468-1253(23)00145-0. Epub 2023 Jun 16. PMID 37336228

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an eosinophilic disorder specialty clinic in the US between April 2018 and January 2020.
Pre-assignment Details: 34 participants screened, 8 excluded (8 did not meet inclusion criteria), and 26 randomized
Groups:
- Benralizumab: Subcutaneous dose of 30 mg of Benralizumab every 4 weeks
  Benralizumab: Benralizumab (anti-IL5Ra) will be injected in doses of 30 mg every 4 weeks (3 times) in subjects with active Eosinophilic Gastritis.
- Placebo: Subcutaneous dose of Placebo every 4 weeks
  Placebo: Placebo will be injected every 4 weeks (3 times) as a comparator to Benralizumab in subjects with active Eosinophilic Gastritis.
Period: Overall Study
Arm/Group | Benralizumab | Placebo
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Benralizumab: Subcutaneous dose of 30 mg of Benralizumab every 4 weeks (total of 3 doses)
- Placebo: Subcutaneous dose of Placebo every 4 weeks (total of 3 doses)
- Total: Total of all reporting groups
Arm/Group | Benralizumab | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (2.0) | 24.1 (7.9) | 19.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
Gastric Peak Eosinophil Count [Median (Inter-Quartile Range); unit: eosinophils per high power field] — Maximum eosinophil count (eosinophils per high power field) in gastric biopsies
  eosinophils per high power field | 210 [93 to 230] | 147 [119 to 208] | 157 [93 to 230]
Gastric Histology Score [Median (Inter-Quartile Range); unit: score on a scale] — Gastric histology score quantifies inflammatory and structural histologic features. Total score is the sum of features scores divided by the maximum possible score. Features include lamina propria eosinophil sheets, periglandular circumferential collars, eosinophils in surface epithelium, eosinophil glandulitis, eosinophil gland abscesses, eosinophils in muscularis mucosa, lamina propria fibroplasia, lamina propria smooth muscle hyperplasia, reactive epithelial changes, acute inflammatory cells, and surface erosion. Scores range from 0 - 1. Higher scores indicate more severe abnormalities.
  score on a scale | 0.55 [0.50 to 0.64] | 0.50 [0.45 to 0.59] | 0.50 [0.45 to 0.64]
Gastric Endoscopy Score (Lanza) [Median (Inter-Quartile Range); unit: score on a scale] — The gastric endoscopy score (Lanza) utilizes standardized criteria for the presence and degree of 5 major endoscopic features (granularity, nodularity, erosion/ulceration, friability, erythema). Total score is the maximum score of the five feature scores from the body, antrum, or fundus. Total scores range from 0 - 14. Higher scores indicate more severe endoscopic findings.
  score on a scale | 4.0 [3.0 to 5.0] | 6.0 [5.0 to 8.0] | 5.0 [4.0 to 6.5]
Blood Eosinophil Count [Median (Inter-Quartile Range); unit: cells per microliter] — Blood absolute eosinophil counts (cell per microliter)
  cells per microliter | 1100 [830 to 2610] | 1640 [710 to 2800] | 1350 [710 to 2630]
SODA Pain Intensity [Median (Inter-Quartile Range); unit: score on a scale] — The symptom of dyspepsia (SODA) questionnaire captures symptoms associated with gastric dyspepsia including symptoms associated with "pain" . Scores range from 0 to 47 for pain. Higher scores indicate more frequent and/or severe symptoms for pain.
  score on a scale | 25 [20 to 30] | 27 [20 to 30] | 26 [20 to 30]
SODA Non-Pain Symptoms [Median (Inter-Quartile Range); unit: score on a scale] — The symptom of dyspepsia (SODA) questionnaire captures symptoms associated with gastric dyspepsia including symptoms associated with "non-pain" . The scores range from 0 to 35 for non-pain. Higher scores indicate more frequent and/or severe symptoms.
  score on a scale | 16 [13 to 17] | 15.5 [13 to 17] | 16 [13 to 17]
SODA Satisfaction [Median (Inter-Quartile Range); unit: score on a scale] — The symptom of dyspepsia (SODA) questionnaire captures general satisfaction associated with present symptoms. The scores range 0 to 23. Higher scores indicate greater Satisfaction.
  score on a scale | 10 [8 to 12] | 8 [4 to 10] | 9 [7 to 11]
EG Diagnostic Panel [Mean (Standard Deviation); unit: delta threshold cycle] — The transcriptomic signature of gastric biopsy samples was obtained using real-time polymerase chain reaction amplification on the Eosinophilic gastritis diagnostic panel (EGDP) comprising a set of 48 gastric transcripts. The EGDP value was calculated by summing the delta CT (threshold cycle) values of the most highly dysregulated genes. Higher values indicate normalization of the transcriptome. Population: Biopsies for gene expression analysis were not collected or failed to yield quality RNA for some subjects
  delta threshold cycle
    number analyzed (Participants) | 9 | 9 | 18
    (all) | -58 (23) | -51 (40) | -55 (32)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients in Histological Remission (<30 Eos/Hpf)
Description: Percent of patients in histologic remission in drug versus placebo groups. Remission is defined as gastric peak eosinophil count < 30 eosinophils per high powered field (eos/hpf).
Time Frame: 12 weeks after start of treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Number; unit: percentage of participants
Groups:
- Benralizumab: Subcutaneous dose of 30 mg of Benralizumab every 4 weeks (total of 3 injections)
- Placebo: Subcutaneous dose of Placebo every 4 weeks (total of 3 injections)
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 13 | 13
percentage of participants | 77 | 8
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Other; p = 0.0001, Fisher Exact

2. Secondary Outcome: Change in Gastric Endoscopic Score (Lanza)
Description: The gastric endoscopic score (Lanza) utilizes standardized criteria for the presence and degree of 5 major endoscopic features (granularity, nodularity, erosion/ulceration, friability, erythema). Total score is the maximum score of the five feature scores from the body, antrum, or fundus. Total scores range from 0 - 14. Change in total endoscopic reference score is defined as post-treatment score minus pre-treatment score. Changes in scores are compared between drug and Placebo. A reduction (negative change) in score indicates improvement.
Time Frame: 12 weeks after start of treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale | -1.0 [-1.0 to 0.0] | 0.0 [-2.0 to 0.0]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Other; p = 0.75, Kruskal-Wallis

3. Secondary Outcome: Change in Gastric Histology Score
Description: The gastric histology score quantifies inflammatory and structural histologic abnormalities in the stomach. Total score is the sum of features scores divided by the maximum possible score for the biopsy. Features include lamina propria eosinophil sheets, periglandular circumferential collars, eosinophils in surface epithelium, eosinophil glandulitis, eosinophil gland abscesses, eosinophils in muscularis mucosa, lamina propria fibroplasia, lamina propria smooth muscle hyperplasia, reactive epithelial changes, acute inflammatory cells, and surface erosion. Total scores range from 0 - 1. Change in gastric total histology scoring is defined as post-treatment total score minus pretreatment total score. Changes in scores are compared between drug and placebo. A reduction (negative change) in score indicates improvement.
Time Frame: 12 weeks after start of treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale | -0.33 [-0.41 to -0.27] | -0.04 [-0.10 to 0.05]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Other; p = 0.006, Kruskal-Wallis

4. Secondary Outcome: Change in Blood Eosinophil Count
Description: Change in absolute eosinophil counts (cells per microliter) is defined as post treatment counts minus pre-treatment counts. Changes in counts are compared between drug and Placebo. A decrease in count is expected due to the effects of the drug.
Time Frame: 12 weeks after start of treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Median (Inter-Quartile Range); unit: cells per microliter
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 13 | 13
cells per microliter | -1060 [-1740 to -830] | -160 [-710 to 120]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Other; p = 0.004, Kruskal-Wallis

5. Secondary Outcome: Change in Eosinophilic Gastritis Diagnostic Panel
Description: The transcriptomic signature of gastric biopsy samples was obtained using real-time polymerase chain reaction amplification on the EG diagnostic panel (EGDP) comprising a set of 48 gastric transcripts. The EGDP value was calculated by summing delta CT (threshold cycle) values of the most highly dysregulated genes. Change is defined as post treatment value minus pre-treatment value. An increase (positive change) indicates improvement (normalization of gene expression).
Time Frame: 12 weeks after start of treatment
Population: Includes participants with pre and post-treatment samples
Measure: Mean (Standard Deviation); unit: delta threshold cycle
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 9 | 9
delta threshold cycle | 29 (31) | -12 (23)
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Other; p = 0.0058, t-test, 2 sided

6. Secondary Outcome: Change in Gastric Peak Eosinophil Count
Description: Change in gastric peak eosinophil count is defined as post-treatment peak count minus pre-treatment peak count. Changes in peak count are compared between Drug and Placebo. A reduction (negative change) in peak count indicates improvement.
Time Frame: 12 weeks after starting treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Median (Inter-Quartile Range); unit: eosinophils per high power field
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 13 | 13
eosinophils per high power field | -132 [-196 to -82] | -29 [-89 to 0]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Test type: Other; p = 0.014, Kruskal-Wallis

7. Secondary Outcome: Change in Clinical Symptoms
Description: The symptom of dyspepsia (SODA) questionnaire captures symptoms associated with gastric dyspepsia including symptoms associated with "pain" and "non-pain" as well as general "satisfaction" with present symptoms. The scores range from 0 to 47 for pain; 0 to 35 for non-pain, and 0 to 23 for satisfaction. Higher scores indicate more frequent and/or severe symptoms for pain and non-pain. Higher scores indicate greater Satisfaction. Change in score is defined as post-treatment total score minus pre-treatment total score. A reduction (negative change) indicates improvement in pain and non-pain. An increase (positive change) indicates improvement in satisfaction.
Time Frame: 12 weeks after start of treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Benralizumab | Placebo
Number analyzed (Participants) | 13 | 13
score on a scale
  Pain score | -3.0 [-9.0 to 0.0] | -2.0 [-6.0 to 0.0]
  Non-pain score | -2.0 [-4.0 to 0.0] | -1.0 [-3.0 to 1.0]
  Satisfaction | 1.0 [0.0 to 5.0] | 2.5 [0.0 to 5.0]
Statistical Analysis 1: Comparison: Benralizumab vs Placebo; Pain Score Comparison; Test type: Other; p = 0.78, Kruskal-Wallis
Statistical Analysis 2: Comparison: Benralizumab vs Placebo; Non-pain score comparison; Test type: Other; p = 0.34, Kruskal-Wallis
Statistical Analysis 3: Comparison: Benralizumab vs Placebo; Satisfaction score comparison; Test type: Other; p = 0.66, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: From informed consent to 4 weeks after the end of the 12 week double-blind. On average, this was approximately 20 weeks.
Arm/Group | Benralizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 11/13 | 8/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Benralizumab (N=13) | Placebo (N=13)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Belching (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Hematochezia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Bacterial overgrowth (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Fever (General disorders) | 2 | 0
Lymphadenopathy (General disorders) | 1 | 0
Sore Throat (General disorders) | 1 | 0
Weight loss (General disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Flu-like Symptoms (Infections and infestations) | 1 | 0
Strep Throat (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 6 | 2
Insomnia (Nervous system disorders) | 0 | 0
Migraine (Nervous system disorders) | 1 | 1
Parasthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT03473977/Prot_SAP_000.pdf